CLINICAL TRIAL: NCT06649942
Title: A Randomized, Single-blind, Placebo-controlled, Four-way Crossover Thorough QT Study to Investigate the Effect of KP-001 on the QT/QTc Interval Using Open-label Moxifloxacin as an Active Control, in Adult Healthy Volunteers
Brief Title: A Study to Evaluate the Effects of KP-001 on the QT/QTc Intervals in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kaken Pharmaceutical (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KP-001-104
Record Dates: First submitted 2024-09-26; First posted 2024-10-21 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers - Male and Female
Keywords: Healty Adults
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment T (Experimental): KP-001 therapeutic dose (KP-001 100 mg + placebo)
  Interventions: Drug: KP-001
- Treatment ST (Experimental): KP-001 supratherapeutic dose (KP-001 400 mg)
  Interventions: Drug: KP-001
- Treatment M (Active Comparator): moxifloxacin 400 mg
  Interventions: Drug: Moxifloxacin 400 mg
- Treatment P (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KP-001 — KP-001 100 mg + placebo
  Arms: Treatment T
Drug: KP-001 — KP-001 400 mg
  Arms: Treatment ST
Drug: Moxifloxacin 400 mg — moxifloxacin 400 mg tablet
  Arms: Treatment M
Drug: Placebo — Placebo
  Arms: Treatment P

SUMMARY:
This is a Phase 1, single-center, randomized, single-blind (participants are blinded), placebo controlled, four-way cross over TQT study (4×4 Williams square design) to investigate the effect of KP-001 on the QTc interval using open-label moxifloxacin as an active control, in adult healthy volunteers.

KP-001 and placebo (dry syrup) will be administered in blinded manner to participants, and the moxifloxacin (tablet) will be administered in open-label manner.Total duration of study participation for each participant is approximately 8 weeks.

Cardiodynamic ECG evaluations will be performed at separate locations and cardiodynamic ECG evaluators will be blinded to treatment group analyzed, ie, blinded to each of the study interventions including moxifloxacin.

DETAILED DESCRIPTION:
This is a Phase 1, single-center, randomized, single-blind (participants are blinded), placebo controlled, four-way cross over TQT study (4×4 Williams square design) to investigate the effect of KP-001 on the QTc interval using open-label moxifloxacin as an active control, in adult healthy volunteers.

KP-001 and placebo (dry syrup) will be administered in blinded manner to participants, and the moxifloxacin (tablet) will be administered in open-label manner.

The study will comprise the following:

* Treatment Periods 1, 2, 3, and 4: For each period, participants will be residential at the Clinical Unit from the day before the dose of study intervention (Day 1 of each treatment period) until 3 days after the dose of study intervention (Day 4 of each treatment period). Participants will receive a single dose of study intervention each period, in accordance with the assigned treatment sequence .
* Washout: at least 7 days between administrations of each study intervention. Total duration of study participation for each participant is approximately 8 weeks.

On Day 1 of Treatment Period 1, participants will be randomly assigned in a 1:1:1:1 ratio to one of the four treatment sequences and administrated a single oral dose of one of the following four treatments under fasting condition:

* KP-001 therapeutic dose (T): KP-001 100 mg + placebo
* KP-001 supratherapeutic dose (ST): KP-001 400 mg
* Placebo (P): placebo dry syrup
* Moxifloxacin (M): moxifloxacin 400 mg tablet

Cardiodynamic ECG evaluations will be performed at separate locations and cardiodynamic ECG evaluators will be blinded to treatment group analyzed, ie, blinded to each of the study interventions including moxifloxacin.

ELIGIBILITY:
Inclusion Criteria:

1. Participant voluntarily agrees to participate in this study and signs an IRB-approved informed consent prior to performing any of the Screening Visit procedures.
2. Males and females between 18 to 55 years of age, inclusive, at the Screening Visit.
3. A female participant is eligible to participate if she is a WONCBP and is not pregnant or breastfeeding.
4. A male participant who is sexually active with female partner(s) of childbearing potential must agree to use both a condom and spermicide from the first dose until 91 days after the last dose of KP-001.
5. A male participant must agree not to donate sperm from the first dose until 91 days after the last dose of KP-001.
6. A continuous nonsmoker who has not used nicotine-containing products for at least 3 months prior to Day -1 of Treatment Period 1 and throughout the study, based on participant self reporting and the result of cotinine test at screening and/or Day -1 of each Treatment Period.
7. Participant is medically healthy with no clinically significant abnormal screening results (eg, medical history, physical examination, laboratory profiles, vital signs, or ECGs), in the opinion of the Investigator or designee. If screening and/or admission results are abnormal, they may be repeated once at screening and/or once at admission to confirm the participant's eligibility.
8. Participant has body weight ≥ 50.0 kg and body mass index within the range 18.0 to 30.0 kg/m2, inclusive, at screening.

Exclusion Criteria:

1. An uninterpretable or abnormal screening and first check-in ECG indicating a second- or third-degree atrioventricular block, or one or more of the following: QRS interval >110 msec; QTcF >450 msec, PR interval >200 msec; HR <40 bpm; T wave abnormalities, or any rhythm other than sinus rhythm that is interpreted by the Principal Investigator and/or qualified designee to be clinically significant.
2. History of risk factors for Torsades de Pointes, including unexplained syncope, known long QT syndrome, heart failure, myocardial infarction, angina, or clinically significant abnormal laboratory assessments including hypokalemia, hypercalcemia, or hypomagnesemia. Participants will also be excluded if there is a family history of long QT syndrome or Brugada syndrome, or family history of sudden cardiac death prior to the age of 40.
3. A sustained supine systolic blood pressure >140 mmHg or <90 mmHg or a supine diastolic blood pressure >90 mmHg or <50 mmHg at screening. A sustained supine systolic blood pressure >150 mmHg or <90 mmHg or a supine diastolic blood pressure >95 mmHg or <50 mmHg at check-in.
4. A resting HR of <40 bpm or >100 bpm when vital signs are measured at screening or check in.
5. Unstable cardiovascular disease, including recent myocardial infarction or cardiac arrhythmia.
6. Participant is legally, mentally or physically incapacitated or, in the opinion of the Investigator, has significant mental or emotional problems, including psychiatric illness (eg, depression and/or anxiety) at the time of the Screening Visit, or that could reasonably be expected to develop during the conduct of the study.
7. Participant has a significant history or clinical manifestation of any metabolic, allergic, dermatologic, hepatic, renal, hematologic, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder as determined by the Investigator or designee.
8. Participant has a history of any illness that, in the opinion of the Investigator or designee, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
9. Participant used any prescription or non-prescription medications (including vitamins, recreational drugs, and dietary or herbal supplements) within 14 days or five half-lives (whichever is longer) prior to Day -1 of Treatment Period 1 and until completion of the Follow-up Call unless, in the opinion of the Investigator, may be treatment for an AE or will not interfere with the interpretation of safety.
10. Participant underwent blood donation or transfusion within 56 days prior to Day -1 of Treatment Period 1 and throughout the study.
11. Participant has a history or presence of hypersensitivity or idiosyncratic reaction to any components of the KP-001 formulation or any components of formulation used as study intervention during the study.
12. Participant has enrolled in a previous clinical study with KP-001 medication.
13. Participant has a history of drug or alcohol abuse (regular alcohol consumption exceeding 14 drinks/week [1 drink = 5 ounces of wine, 12 ounces of beer, or 1.5 ounces of hard liquor] within one year before the Screening Visit).
14. Participant has a complication of drug allergies or history of drug allergies.
15. Participant used any investigational drug in the last 30 days or five half-lives (if known), whichever is longer, prior to Day -1 of Treatment Period 1.
16. Participant had any major illness within 30 days before the Screening Visit.
17. Participant had any major surgical procedure within 30 days prior to Day -1 of Treatment Period 1 or any planned surgery during study period.
18. Participant had any laboratory abnormality that, in the judgment of the Investigator, would put the participant at unacceptable risk for participation in the study or may interfere with the assessments included in the study.
19. Participant has abnormal findings on the screening ECG deemed clinically significant by the Investigator or qualified designee.
20. Participant is an employee of the Sponsor or any CRO involved in the study, the Investigator, or an immediate family member (partner, offspring, parents, siblings, or sibling's offspring) of an employee involved in the study.
21. Participant has consumed alcohol- or caffeine-containing foods and beverages within 72 hours prior to Day -1 of Treatment Period 1 and does not agree to refrain from consuming during the entire study, unless deemed acceptable by the Investigator.
22. Participant has positive urine drug or urine alcohol and positive cotinine test results at screening or Day -1 of Treatment Period 1.
23. Participant has consumed grapefruit-containing foods and beverages within 7 days prior to Day -1 of Treatment Period 1 and does not agree to refrain from consuming during the entire study.
24. Participant has consumed St. John's wort-containing foods and beverages within 14 days prior to Day -1 of Treatment Period 1 and does not agree to refrain from consuming during the entire study.
25. Participant is unable or unwilling to undergo multiple venipunctures.
26. Participant has a history or presence of liver disease or cholecystectomy within one year prior to screening.
27. Participant has an HbA1c >5.7% at screening.
28. Participant has positive results at screening for human immunodeficiency virus, hepatitis B core antibody, hepatitis B surface antigen or hepatitis C virus.
29. Participant has a disorder or any condition that would interfere with the absorption, distribution, metabolism, or excretion of drugs.
30. Participant has eGFR calculated using the CKD-EPI formula <80 mL/min at screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Largest time-matched placebo-corrected change from baseline in QTcF (ΔΔQTcF) collected in a 24-hour period after KP-001 single dosing | Before dosing (Baseline) through 24 hours
  To evaluate the effect of KP-001 as single therapeutic and supratherapeutic dose on the QTcF interval

SECONDARY OUTCOMES:
Placebo-corrected change from baseline in QTcF (ΔΔQTcF) | Before dosing (Baseline) through 24 hours
  To study the concentration-response relationship between KP-001 concentrations after dosing and ΔQTcF (C-ΔQTcF model)
Largest time-matched placebo-corrected change from baseline in QTcF (ΔΔQTcF) after moxifloxacin dosing | Before dosing (Baseline) through 24 hours
  Largest time-matched placebo-corrected change from baseline in QTcF (ΔΔQTcF) collected in a 24-hour period after moxifloxacin dosing
Categorial outliers for QRS after KP-001 dosing | Before dosing (Baseline) through 24 hours
Placebo-corrected ΔHR after KP-001 dosing | Before dosing (Baseline) through 24 hours
Placebo-corrected ΔPR after KP-001 dosing | Before dosing (Baseline) through 24 hours
Placebo-corrected ΔQRS after KP-001 dosing | Before dosing (Baseline) through 24 hours
Categorial outliers for PR after KP-001 dosing | Before dosing (Baseline) through 24 hours
Categorial outliers for HR after KP-001 dosing | Before dosing (Baseline) through 24 hours
Categorial outliers for QTcF after KP-001 dosing | Before dosing (Baseline) through 24 hours
Change from baseline PR after KP-001 dosing | Before dosing (Baseline) through 24 hours
Change from baseline HR after KP-001 dosing | Before dosing (Baseline) through 24 hours
PK parameters of KP-001 in plasma: CLtot/F | pre-dose and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 36 and 72 hours post-dose
PK parameters of KP-001 in plasma: Tmax | pre-dose and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose
  To evaluate PK of KP-001
PK parameters of KP-001 in plasma: t1/2 | pre-dose and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose
  To evaluate PK of KP-001
PK parameters of KP-001 in plasma: Vz/F | pre-dose and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose
  To evaluate PK of KP-001
Frequency of treatment-emergent morphology and appearance of U-wave after KP-001 dosing | Before dosing (Baseline) through 24 hours
PK parameters of KP-001 in plasma: Cmax | pre-dose and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose
  To evaluate PK of KP-001
Frequency of treatment-emergent changes in Twave morphology after KP-001 dosing | Before dosing (Baseline) through 24 hours
PK parameters of KP-001 in plasma: AUC0-24 | pre-dose and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose
PK parameters of KP-001 in plasma: AUC0-48 | pre-dose and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose
PK parameters of KP-001 in plasma: AUC0-72 | pre-dose and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose
PK parameters of KP-001 in plasma: AUCinf | pre-dose and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose
  Area Under the Concentration Time-curve From Time Zero to Infinity for KP-001
Placebo-corrected change from baseline in QTcF (ΔΔQTcF) predicted from the C-ΔQTcF model at Cmax | Before dosing (Baseline) through 24 hours
  To study the concentration-response relationship between KP-001 concentrations

CONTACTS AND LOCATIONS:
Locations (1):
- Parexel Early Phase Clinical Unit - Los Angeles, Glendale, California, United States